CLINICAL TRIAL: NCT02154893
Title: Synergic Effects of Ultrasound and Laser on the Pain Relief and Functionality in Women With Hand or Knee Osteoarthritis.
Brief Title: Synergic Effects of Ultrasound and Laser on the Pain Relief and Functionality
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fernanda Rossi Paolillo, Ph.D, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP2013
Record Dates: First submitted 2014-05-24; First posted 2014-06-03 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2014-05

CONDITIONS: Osteoarthritis
Keywords: Ultrasound; Laser; Therapeutic exercise; Rehabilitation; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Ultrasonography; Lasers; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Device and exercise (Experimental): Device with ultrasound and laser associated with therapeutic exercise
  Interventions: Device: Ultrasound plus Laser and therapeutic exercise
- Device (Experimental): Device with ultrasound and laser
  Interventions: Device: Ultrasound plus Laser
- Placebo (Placebo Comparator): Without any treatment
  Interventions: Device: Utrasound plus Laser Placebo

INTERVENTIONS:
Device: Ultrasound plus Laser and therapeutic exercise — Ultrasound with frequency 1 Mhz and infrared laser with output power at 100 mW. The resistance training was performed.The treatments are done once a week, for 3 months.
  Arms: Device and exercise
Device: Ultrasound plus Laser — Ultrasound with frequency 1 Mhz and infrared laser with output power at 100 mW. The treatments are done once a week, for 3 months.
  Arms: Device
Device: Utrasound plus Laser Placebo — The device with Ultrasound and infrared laser without emitting electromagnetic or mechanical waves was applied (null dose).
  Arms: Placebo

SUMMARY:
There are several therapeutic effects of the ultrasound (US) or low level laser therapy (LLLT), including pain relief, increase of microcirculation, modulation of inflammatory response and accelerated tissue repair. The investigators hypothesis was that a combination of US, LLLT and therapeutic exercise may maximize clinical outcome.

DETAILED DESCRIPTION:
Patients with pain, especially chronic pain, avoid movements. This is turn results in a gradual impairment of their physical condition, reducing, for example, strength, flexibility, physical functionality and occupational activity. To performed physical treatments, a prototype device was development. The device includes four diode laser beams (808 nm) around of the one ultrasound transducer.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian women
* Aged between 60 and 80 years
* Hand osteoarthritis
* Knee osteoarthritis

Exclusion Criteria:

* Psychiatric disorder,
* Neurological disease
* Metabolic disease
* Pulmonary disease
* Cardiac disease,
* Thrombosis
* Cancer.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Analysis of pain for hands and knees | 3 months
  Pressure pain thresholds by algometry (N)

SECONDARY OUTCOMES:
Subjective pain scale for hands and knees | 3 months
  Pain intensity by visual analog scale (VAS)
Jebsen-Taylor Hand Function Test | 3 months
  The time (s) to perform different activities is registered
Box and block Hand Function Test | 3 months
  The number of wooden blocks that can be transported from one compartement of a box to another within 1 min is counted
Toe-Touching Function Test | 3 months
  The distance (cm) from the finger of hand to finger of foot is registered
Sit-to-Stand Function Test | 3 months
  The number of sit-to-stand within 1 min is counted
Gait Function Test | 3 months
  The time (s) to perform 10 meters walked is registered
Balance Function Test | 3 months
  The time (s) to perform static and dynamic balance is registered
Dynamometry | 3 months
  Strength (N)
Accelerometer | 3 months
  Acceleration (km.h-1)
Electrogoniometry | 3 months
  Range of motion (angle)
Quality of life Questionnaire | 3 months
  SF36
Questionnaire for Osteoarthritis | 3 months
  AUSCAN, WOMAC, KOOS, LEQUESNE index

CONTACTS AND LOCATIONS:
Overall Officials: Vanderlei S Bagnato, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Alessandra R Paolillo, Ph.D, Study Director — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Fernanda R Paolillo, Ph.D, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Jéssica João, PT, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP); Herbert João, Msc, Principal Investigator — Physics Institute of São Carlos (IFSC), University of São Paulo (USP)
Locations (1):
- Alessandra Rossi Paolillo, São Carlos, São Paulo, Brazil

REFERENCES:
- [Result] Brosseau L, Wells G, Marchand S, Gaboury I, Stokes B, Morin M, Casimiro L, Yonge K, Tugwell P. Randomized controlled trial on low level laser therapy (LLLT) in the treatment of osteoarthritis (OA) of the hand. Lasers Surg Med. 2005 Mar;36(3):210-9. doi: 10.1002/lsm.20137. PMID 15704096
- [Result] Ekim A, Armagan O, Tascioglu F, Oner C, Colak M. Effect of low level laser therapy in rheumatoid arthritis patients with carpal tunnel syndrome. Swiss Med Wkly. 2007 Jun 16;137(23-24):347-52. doi: 10.4414/smw.2007.11581. PMID 17629805
- [Result] Allen RJ. Physical agents used in the management of chronic pain by physical therapists. Phys Med Rehabil Clin N Am. 2006 May;17(2):315-45. doi: 10.1016/j.pmr.2005.12.007. PMID 16616270
- [Result] Korstjens CM, van der Rijt RH, Albers GH, Semeins CM, Klein-Nulend J. Low-intensity pulsed ultrasound affects human articular chondrocytes in vitro. Med Biol Eng Comput. 2008 Dec;46(12):1263-70. doi: 10.1007/s11517-008-0409-9. Epub 2008 Oct 14. PMID 18853213
- [Result] Tascioglu F, Kuzgun S, Armagan O, Ogutler G. Short-term effectiveness of ultrasound therapy in knee osteoarthritis. J Int Med Res. 2010 Jul-Aug;38(4):1233-42. doi: 10.1177/147323001003800404. PMID 20925995
- See also: Optics and Photonics Research Center — http://cepof.ifsc.usp.br/